CLINICAL TRIAL: NCT05659888
Title: PENELOPE-CTRL: Real Life Lipid Management Compared to Protocolized Implementation of the Current Dutch- and ESC-guidelines in Very High-risk CV-patients
Brief Title: Real Life Lipid Management in Hospitals Not Participating in PENELOPE Trial - Control Population for PENELOPE
Acronym: PENELOPECTRL
Status: Completed | Type: Observational
Sponsor: Clinical Operations WCN B.V. (Network)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: DCV-2017-11843
Record Dates: First submitted 2022-12-12; First posted 2022-12-21 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Atherosclerotic Cardiovascular Disease; STEMI; Non STEMI
MeSH Terms: conditions — Atherosclerosis; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Guideline recommended evidence-based clinical care correlates with improved patient outcomes. In real life care, however, adherence to guideline recommendations remains suboptimal. In real life, patients may receive suboptimal treatment and as a result treatment targets are not always met. To support and improve secondary prevention for cardiovascular disease, PENELOPE and PENELOPE-CTRL are designed to support guideline implementation on lipid management and provide valuable feedback to care-givers on real world data.

DETAILED DESCRIPTION:
The recent PENELOPE study was designed to determine the effect of a protocolized, Dutch-, and ESC- guideline based strategy of stepwise intensified lipid management in patients at very high risk for ACS. In PENELOPE 22 Dutch non-academic hospitals, members of the WCN investigator network, implemented a protocol guided guideline approach in a consecutive cohort of very high-risk patients admitted for ACS over the period 01-01-2019 to 31-08-2020. Lipid values and medication strategy are collected at baseline (index ACS), and after three months and one year post ACS, in order to establish the percentage of patients on target (LDL).

The current PENELOPE-CTRL study on the other hand, is designed to serve as a contemporary control cohort for PENELOPE. PENELOPE-CTRL is a retrospective observational study, creating a contemporary snapshot of real-life lipid management for secondary prevention in very high-risk patients. PENELOPE-CTRL will collect data in similar hospitals who did not participate in the PENELOPE trial.

To allow comparison of these two strategies, protocol guided versus real life implementation of the cholesterol treatment guidelines, both cohorts include similar patients, and similar data will be collected (e.g., lipid lowering drugs, lipid panels) . Analysis will be done at similar time points.

Comparing the real-life data from PENELOPE-CTRL with the data from the PENELOPE study will quantify the effect of a strategy of protocolized guideline-based lipid management with regards to the incidence of target LDL-C levels in very high-risk patients, 3 months and one year after hospitalisation with a myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 and ≤70 years
* Alive at hospital discharge after admission for (N)STEMI between 1-1-2019 and 31-08-2020
* Planned for follow-up at a participating PENELOPE CTRL site
* History of T2DM and/or history of ASCVD defined as either one of:

  * cerebrovascular disease/ event: transient ischemic attack, cerebral infarction, amaurosis fugax, retinal infarction
  * Coronary artery disease/ event: unstable angina pectoris, MI, ACS, coronary revascularization (coronary angioplasty or surgical procedure for coronary bypass)
  * Peripheral artery disease (symptomatic and documented obstruction of a distal extremity artery or surgical intervention (percutaneous transluminal angioplasty, bypass or amputation)

Exclusion Criteria:

* Pregnant and lactating women
* Participation in lipid modifying drug trials up to two years after index cardiovascular event

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a history of ASCVD and/or type 2 diabetes (T2DM), admitted for a type I ST-elevation myocardial infarct (STEMI) or non-STEMI. Patients <18 years or >70 years of age will be excluded.
  In PENELOPE patients over 70 were included based on a frailty index. As this parameter cannot be determined retrospectively, patients over 70 will be excluded from the CTRL cohort, as well as from the comparative analysis for the two cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 827 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients reaching the LDL-C target level (≤ 1.8 mmol/L) | 3 months
  reaching LDL-C target level (≤ 1.8 mmol/L) 3 months after admission for a type I (N)STEMI, compared to the designated PENELOPE cohort

SECONDARY OUTCOMES:
Incidence of LDL-C target level (≤ 1.8 mmol/L) | 1 year
  Incidence of LDL-C (≤ 1.8 mmol/L) at baseline (admission for a type I (N)STEMI), 3 months and 1 year after baseline, compared to the designated PENELOPE cohort.
Incidence of LDL-C target level (≤ 1.4 mmol/L) | 1 year
  Incidence of LDL-C (≤ 1.4 mmol/L) at baseline (admission for a type I (N)STEMI), 3 months and 1 year after baseline, compared to the designated PENELOPE cohort.
incidence of achieving 50% LDL-C reduction | 1 year
  Incidence of achieving 50% LDL-C reduction compared to baseline, after 3 months and 1 year, also adjusted to the start date of the related drug regimen.
LLT compared to PENELOPE cohort | 1 year
  Lipid lowering therapy at baseline, after 3 months and 1 year, compared to the designated PENELOPE cohort.
LDL-C level 3 months after adjustment | 3 months
  LDL-C level at 3 months, also adjusted to the start date of the related drug regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Alings, Principal Investigator — WCN
Locations (13):
- Netherlands (13):
  - NoordWest Hospital (NWZ), Alkmaar
  - Reinier de Graaf Hospital, Delft
  - Deventer Hospital, Deventer
  - Treant Hospital, Emmen
  - Saxenburg Medisch Centrum, Hardenberg
  - Elkerliek Hospital, Helmond
  - Alrijne Hospital, Leiden
  - Isala Hospital, Meppel
  - Canisius Wilhemina Hospital (CWZ), Nijmegen
  - Haaglanden Hospital, The Hague
  - Haga Hospital, The Hague
  - Diakonessenhuis Utrecht, Utrecht
  - Maxima Medisch Centrum, Veldhoven

DOCUMENTS (1):
  • Study Protocol (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT05659888/Prot_001.pdf